CLINICAL TRIAL: NCT00173836
Title: Swallowing Pattern of Patients With Nasopharyngeal Cancer Before and After Radiation Therapy: Longitudinal Study and Correction With Saliva Amount
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yeun-Chung Chang, National Taiwan University Hospital
Other Study IDs: Yeun-Chung Chang; NSC 92-2218-E-227-001
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2009-09-09 (Estimated); Status verified 2009-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; Saliva; Swallowing; Videofluoroscopy; Radiation
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Significant evidence has shown that radiation therapy for patients with nasopharyngeal cancer (NPC) can cause swallowing abnormality. Based on our prior cross-sectional study for 184 NPC patients from 1995 to 1999, the findings of videofluoroscopic swallowing study (VFSS) revealed continuous deterioration of swallowing function of these patients even many years after radiation. We conducted a prospective study to evaluate the longitudinal change of swallowing function based on VFSS before, one month, one year and two years after completing radiation therapy. The amount of saliva was measured at the same time of VFSS study to test the relationship of decreased amount of saliva and swallowing function. Comparison of serial VFSS studies in NPC patients (n=84) and normal volunteers (n=38) were obtained. We assume that this study may reveal a complete understanding of changing swallowing patterns in the course of radiation therapy of patients with NPC. From this study, NPC patients can understand their own swallowing function. Therefore, the information may enable for earlier intervention of swallowing training or correction to avoid morbidity of radiation therapy in this patient group.

ELIGIBILITY:
Inclusion Criteria:

Nasopharyngeal cancer patients > 20 yrs.

Exclusion Criteria:

pregnant women

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nasopharyngeal cancer patients
Sampling Method: Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2003-08; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yeun-Chung Chang, M.D., Ph.D., Principal Investigator — National Taiwan Univserity Hospital and College of Medicine
Locations (1):
- X-ray fluoroscopy, Taipei, Taiwan

REFERENCES:
- [Background] Chang YC, Chen SY, Lui LT, Wang TG, Wang TC, Hsiao TY, Li YW, Lien IN. Dysphagia in patients with nasopharyngeal cancer after radiation therapy: a videofluoroscopic swallowing study. Dysphagia. 2003 Spring;18(2):135-43. doi: 10.1007/s00455-002-0096-x. PMID 12825907